CLINICAL TRIAL: NCT01866826
Title: A Double Blind Randomized Placebo Controlled Study Examining the Effects of a Non-Absorbable (Rifaximin) Antibiotic on the Chronic Immune Activation Observed In HIV-infected Subjects
Brief Title: Rifaximin for Chronic Immune Activation in People With HIV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Pittsburgh (Other); Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Frank Maldarelli, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 130062; 13-I-0062 (Other: NIAID)
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: HIV
Keywords: HIV; Eradication Strategies; Immune Activation
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIV Infected Subjects (Experimental): Human immunodeficiency virus (HIV) infected subjects with viral suppression on antiretroviral (ART). Double-blinded/placebo controlled trial with cross-over design. Rifaximin
  Interventions: Drug: Rifaximin
- HIV Infected Subjects Placebo (Placebo Comparator): HIV infected subjects with viral suppression on ART. Double-blinded/placebo controlled trial with cross-over design. Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rifaximin — subject will receive three capsules of rifaximin (183.3 mg each) by mouth twice daily (total 1100 mg Daily)
  Other Names: Xifaxan
  Arms: HIV Infected Subjects
Other: Placebo — subject will receive three capsules of placebo by mouth twice daily.
  Arms: HIV Infected Subjects Placebo

SUMMARY:
Background:

* Human immunodeficiency virus (HIV) treatment can control the amount of virus in the blood, but it does not provide a cure. The reasons why HIV treatment does not cure the infection are not well understood. HIV persists in blood cells for years, even if people receive treatment for it. In addition, HIV infection leads to an activated immune system, which can cause other problems.
* One theory for why HIV infection causes immune activation involves the intestinal tract. HIV infects immune cells the intestine soon after infection and damages their immune barrier. This damage lets bacteria cross into the bloodstream, leading to ongoing inflammation. Even when a person with HIV feels well, this chronic inflammation may affect the immune system. Researchers want to see if the antibiotic Rifaximin can reduce this inflammation. Rifaximin is designed to stay inside the digestive system, so it affects only bacteria in the intestines.

Objectives:

- To see if Rifaximin can reduce bacteria-related inflammation in people with HIV.

Eligibility:

- Individuals at least 18 years of age who have HIV infection and are taking medications to treat it.

Design:

* Participants will be screened with a physical exam, blood test, and medical history.
* Participants will take either Rifaximin or a placebo for 4 weeks. They will have no medication for 4 to 6 weeks, and then take the other drug for 4 more weeks.
* During the study, participants will have frequent blood and urine tests. They will also provide stool samples. Liver and kidney function tests will be performed. HIV viral load (the amount of virus in the blood) will also be studied.
* Participants will have a final follow-up visit after an additional 4 weeks.
* Two additional tests are optional for study participants:
* Two blood draws: one on the third day after starting Rifaximin, and one on the third day after starting the placebo.
* Up to three colonoscopies of the lower intestine and biopsies of the intestine. These studies will collect samples of the intestinal tract to look at the effects of Rifaximin in the study.

DETAILED DESCRIPTION:
The introduction of antiretroviral therapy (ART) has resulted in dramatic reductions in acquired immune deficiency syndrome (AIDS) related morbidity and mortality. Therapy is not curative, however, and the nature of human immunodeficiency virus (HIV) replication during therapy remains unclear. Understanding mechanisms involved in HIV persistence will be useful in identifying effective strategies for HIV eradication. Immune activation (IA) plays a central role in the pathogenesis of HIV-infection, and may play a critical role in HIV persistence during therapy. In comparison with the levels detected in HIV uninfected subjects, both cellular markers of activation and biomarkers of inflammation are elevated in HIV-infected individuals. Levels of inflammatory cytokines and cellular markers of activation independently correlate with disease progression in HIV-infected subjects. Chronic, persistent IA is associated with the observed cluster of differentiation (CD4) depletion in untreated subjects and among ART- treated and virologically suppressed subjects and may contribute to the failure to reconstitute CD4 counts. IA also plays a role in the pathogenesis of non-AIDS related complications such as chronic kidney and coronary artery disease (CAD).

Although chronic persistent IA may play a role in HIV persistence, the source of immune activation itself is unknown. Low level viremia may represent a virologic stimulus for IA. Viremia persists at low levels during therapy, but it is not known whether HIV infection is maintained by ongoing cycles of replication in sanctuary sites, production from long-lived cells with integrated proviruses, or both. Using sensitive assays for HIV-1 viremia, we and others have detected the presence of persistent HIV viremia in the majority of subjects throughout prolonged antiretroviral therapy. Drug intensification studies suggest little contribution of active replication to levels of persistent viremia, suggesting that factors other than complete cycles of HIV replication may contribute to HIV-1 persistence. Activation of HIV-1 from long-lived cells in reservoir sites is another potential source of viremia, but the nature of such reservoirs is not yet well understood.

The mechanism of immune activation in HIV infection remains to be clarified and is likely multifactorial. Additional potential mechanisms of persistence include a central role for the gastrointestinal tract. The gastrointestinal epithelium and gut-associated lymphoid tissue (GALT) are thought to represent important barriers to microbial translocation, but HIV infection results in substantial destruction of both barriers. The reservoir of bacteria in the gastrointestinal tract is substantial, and small amounts of bacterial products are reported to translocate across the gastrointestinal tract into the bloodstream; microbial translocation across this defective GALT is an important driver of the observed immune activation in HIV infection. The precise effects of ART on gut microbial translocation remain uncertain; some studies suggest that ART incompletely reverses the effects of microbial translocation, others have failed to demonstrate any effect, yet other studies have demonstrated complete reversal with ART.

In this study, we will examine the potential role of bacterial translocation on IA by studying the effects of the antibiotic rifaximin on markers of microbial translocation, immune activation, and HIV viremia in the gut reservoir in ART treated aviremic subjects. Rifaximin is an orally administered antibiotic with potent qualitative and quantitative effects on gut bacterial flora. Rifaximin is not systemically absorbed, and drug effects appear to be confined to the gastrointestinal tract. Rifaximin has been studied as maintenance therapy in both inflammatory bowel disease (IBD) and hepatic encephalopathy (HE), disease states in which endogenous gut flora play an important role in the pathogenesis. It is anticipated that the use of rifaximin will result in an alteration and reduction in gut bacterial flora. We hypothesize that the reductions in gut bacterial flora will result in a corresponding reduction in bacterial translocation and reductions in biologically active lipopolysaccharides (LPS) levels leading to reductions in immune aced persons receiving Activation, and HIV.

In this protocol, the role of gut microbial translocation in the pathogenesis of HIV infection will be examined by performing a randomized, double-blind, placebo-controlled study of rifaximin with a case cross-over design in virologically-suppressed HIV-infected persons receiving ART.

ELIGIBILITY:
* PARTICIPANT INCLUSION CRITERIA:

Patients who have agreed in the course of other research studies to have their records reviewed will have the following elements evaluated from their existing records: age, history of human immunodeficiency virus (HIV) infection, antiretroviral therapy (ART) history and viral loads prior to informed consent, or else these elements will be assessed after informed consent. All blood draws to assess eligibility will be completed after obtaining informed consent. To participate in this study the criteria listed below will need to be met.

1. Subjects must be 18 years of age or older.
2. Able and willing to provide written informed consent
3. Must have a history of documented HIV infection.
4. HIV infection if not previously documented at host institutions will need to be documented by a plasma human immunodeficiency virus (HIV) ribonucleic acid (RNA) viral load, rapid HIV test or any other licensed enzyme-linked immunosorbent assay (ELISA) test and confirmed by another test using a different method such as a rapid HIV test, Western Blot, HIV culture, HIV antigen, HIV pro-viral deoxyribonucleic acid (DNA) at any time prior to study entry.
5. ART- treated subjects who are virologically suppressed for greater than or equal to 3 years (1095 days). To meet this criteria all documented viral loads in the 3 years (1095 days) prior to the screening visit must be below the lower limit of detection [LLD] using Food and Drug Administration (FDA)-approved standard assays (i.e. <50 copies/mL) with the following clarification: In each of the three prior years, subjects experiencing a single blip [i.e. viral loads above the lower limit of detection, LLD] may be included provided they satisfy the following criteria: the blips are below 200 copies/ml, and the blip is surrounded (i.e the preceding and succeeding viral loads) by undetectable HIV-1 RNA level measurements. That is all viral loads must be below LLD EXCEPT for up to one blip. In any 12 month period.
6. Viral RNA level < 50 c/ml at Screen 1.
7. A minimum of 2 HIV-1 RNA levels that are below the lower limit of detection using standard assays will be required during the 12 month period prior to their screening visit. As assay characteristics across the sites can vary, LLD for the assay will be used to define whether or not a subject is suppressed.
8. Stable dose of statin therapy for 6 months if receiving statin therapy.
9. No known allergy or contraindication to the use of rifamycin compounds such as rifampin, rifabutin or rifaximin. .
10. The effect of rifaximin on the developing human fetus are unknown, therefore subjects must be willing to use two methods of contraception (one of which must be a barrier method) during the study period. Adequate methods of birth control include: tubal ligation, hysterectomy, condoms (male or female) with or without a spermicide; diaphragm or cervical cap with spermicide; intrauterine device; any of the methods that require a prescription (such as contraceptive pills or patch, Norplant, Depo-Provera, and others) or a male partner who has previously undergone a vasectomy.

The following elements will be assessed with a blood draw and after obtaining informed consent.

1. Absolute Neutrophil count (ANC) greater than or equal to 750/mm(3)
2. Hemoglobin greater than or equal to 10.0 g/dL for women and Hemoglobin 11.0 g/dl for men
3. Platelet count greater than or equal to 75,000/mm(3)
4. Estimated Glomerular Filtration Rate (eGFR) >60 mL/min, eGFR will be calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
5. Confirmed serum glutamate pyruvate transaminase (SGPT)/serum glutamate oxaloacetate transferase (SGOT) less than or equal to 3 times the upper limit of normal (ULN)
6. International Normalized Ratio (INR) less than or equal to the upper limit of normal (ULN) for the assay
7. Negative urine pregnancy test of child bearing potential at randomization
8. No evidence of active hepatitis B or hepatitis C (active hepatitis B will be defined as a positive hepatitis B surface antigen present on a single determination, whereas a positive result on hepatitis C RNA will be considered as evidence of active hepatitis C)

All routine laboratory testing used to determine safety will be completed within the 70 days prior to randomization.

EXCLUSION CRITERIA:

1. Known bleeding diathesis (for example a diagnosis of hemophilia or Von Willebrand disease)
2. Active drug use or alcohol abuse/dependence, which in the opinion of the investigators will interfere with the patients ability to participate in the study
3. Serious illness requiring systemic treatment and/or hospitalization within 30 days of screening into the study
4. Evidence of active opportunistic infections or neoplasms (excluding cutaneous basal cell carcinoma and squamous cell carcinoma) in the 6 months prior to randomization
5. History of inflammatory bowel disease (Crohn's Disease, ulcerative colitis)
6. Positive urine pregnancy test at screening (of child bearing potential).
7. Breastfeeding
8. Current imprisonment
9. Concurrent immunomodulatory agents, including systemic corticosteroids in the 12 weeks prior to randomization. Topical, nasal or inhaled corticosteroid use is allowed
10. Concomitant use of probiotics except yogurt
11. Chronic antibiotic use such as tetracyclines for acne
12. Vaccinations within 6 weeks of randomization
13. Concomitant use of anticoagulants (other than aspirin and nonsteroidal anti-inflammatory drugs (NSAIDS)) is an exclusion criterion for subjects opting in for the colonoscopy. Aspirin and NSAIDs will be discontinued per each institutions requirement before the procedure.
14. Child-Pugh Class C disease
15. A prior history of Clostridium difficile colitis
16. Any condition that precludes the safe administration of conscious sedation for endoscopy (such as decompensated lung or heart disease) will not be able to participate in the colonoscopy aspect of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-01-18 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Maldarelli, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - Walter Reed National Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deeks SG. Immune dysfunction, inflammation, and accelerated aging in patients on antiretroviral therapy. Top HIV Med. 2009 Sep-Oct;17(4):118-23. PMID 19890183
- [Background] Kuller LH, Tracy R, Belloso W, De Wit S, Drummond F, Lane HC, Ledergerber B, Lundgren J, Neuhaus J, Nixon D, Paton NI, Neaton JD; INSIGHT SMART Study Group. Inflammatory and coagulation biomarkers and mortality in patients with HIV infection. PLoS Med. 2008 Oct 21;5(10):e203. doi: 10.1371/journal.pmed.0050203. PMID 18942885
- [Background] Hunt PW, Martin JN, Sinclair E, Bredt B, Hagos E, Lampiris H, Deeks SG. T cell activation is associated with lower CD4+ T cell gains in human immunodeficiency virus-infected patients with sustained viral suppression during antiretroviral therapy. J Infect Dis. 2003 May 15;187(10):1534-43. doi: 10.1086/374786. Epub 2003 Apr 23. PMID 12721933
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-I-0062.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Upon completion of a 4 week course of rifaximin or placebo subjects will undergo a 4-6 week washout period and cross over treatment assignments to complete a 4 week course of either rifaximin or placebo.
Groups:
- Rifaximin, Then Placebo: Human immunodeficiency virus (HIV) infected subjects with viral suppression on antiretroviral (ART). Double-blinded/placebo controlled trial with cross-over design.
  Subject will receive three capsules of rifaximin (183.3 mg each) by mouth twice daily (total 1100 mg Daily) for 4 weeks, followed by a 4-6 week washout period, and then will receive three capsules of placebo by mouth twice daily for 4 weeks.
- Placebo, Then Rifaximin: HIV infected subjects with viral suppression on ART. Double-blinded/placebo controlled trial with cross-over design. Placebo
  Subject will receive three capsules of placebo by mouth twice daily for 4 weeks, followed by a 4-6 week washout period, and then will receive three capsules of rifaximin (183.3 mg each) by mouth twice daily (total 1100 mg Daily) for 4 weeks.
Period: Phase I -Initial Randomization - 4 Weeks
Arm/Group | Rifaximin, Then Placebo | Placebo, Then Rifaximin
Started | 23 | 23
Completed | 22 | 23
Not Completed | 1 | 0
Not completed — Post Enrollment Withdrawal | 1 | 0
Period: Wash-Out Period - 4 -6 Weeks
Arm/Group | Rifaximin, Then Placebo | Placebo, Then Rifaximin
Started | 22 | 23
Completed | 22 | 20
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Post Enrollment Withdrawal | 0 | 1
Period: Second Intervention - 4 Weeks
Arm/Group | Rifaximin, Then Placebo | Placebo, Then Rifaximin
Started | 22 | 20
Completed | 22 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All human immunodeficiency virus (HIV) infected subjects with viral suppression on antiretroviral (ART). Double-blinded/placebo controlled trial with cross-over design.
Arm/Group | All Participants
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.609 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 25
  More than one race | 1
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Changes in Soluble Cluster of Differentiation 14 (sCD14) Levels Between the Placebo and Rifaximin Phases of the Study
Description: One sample Wilcoxon statistic was applied to evaluate the difference on treatment phases between the placebo and Rifaximin.
Time Frame: Between Day 28 of Treatment Phase 1 and Day 28 of Treatment Phase 2
Population: 46 randomized participants, 37 had evaluable results. Number of participants analyzed differ from Participant Flow because it represents the cumulative number of participants analyzed per Arm/Group for this outcome measure.
Measure: Mean (Inter-Quartile Range); unit: mcg/mL
Groups:
- Rifaximin: Human immunodeficiency virus (HIV) infected subjects with viral suppression on antiretroviral (ART). Double-blinded/placebo controlled trial with cross-over design.
  Rifaximim: subject will receive three capsules of rifaximin (183.3 mg each) by mouth twice daily (total 1100 mg Daily).
- Placebo: HIV infected subjects with viral suppression on ART. Double-blinded/placebo controlled trial with cross-over design.
  Placebo: Subject will receive three capsules of placebo by mouth twice daily.
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 37 | 37
mcg/mL | 0.0067 [-0.0097 to 0.22] | 0.0035 [-0.195 to 0.154]
Statistical Analysis 1: Comparison: Rifaximin vs Placebo; Test type: Superiority; p = 0.51, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Participants With Viral (HIV-1)-Ribonucleic Acid (RNA) Elevated by Greater Than 50 Copies/ml Plasma at the End of the Rifaximin or Placebo Phase
Description: HIV-1-RNA levels were assessed by using the single copy assay or the traditional HIV Branched Deoxyribonucleic Acid bDNA assay to determine elevations in HIV-1 RNA >50 copies/ml plasma at the end of the Rifaximin or placebo phase. Differences were tested by using both the Wilcoxon and the t-test.
Time Frame: Between Day 28 of Treatment Phase 1 and Day 28 of Treatment Phase 2
Population: Number of participants analyzed differ from Participant Flow because it represents the cumulative number of participants analyzed per Arm/Group for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 43 | 43
Participants | 0 | 0
Statistical Analysis 1: Comparison: Rifaximin vs Placebo; We calculated the proportion of pts with elevated viral levels >50 copies/ml at each phase of the study; Test type: Superiority; We estimated that four of the seven patients would have an elevation in viral Ribonucleic Acid (RNA) level >50 copies/ml

3. Secondary Outcome: Changes in Soluble Markers of Inflammation Between the Placebo and Rifaximin Phases of the Study
Description: Changes in soluble marker of inflammation Interleukin 6 (IL6) between the placebo and rifaximin phases of the study. Differences will be tested by using both the Wilcoxon and the t-test.
Time Frame: Between Day 28 of Treatment Phase 1 and Day 28 of Treatment Phase 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: picograms/milliliter
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 37 | 37
picograms/milliliter | 7.94 (3.89) | 8.10 (3.70)

4. Secondary Outcome: Changes in Cellular Markers of Immune Activation Between the Placebo and Rifaximin Phases of the Study
Description: Changes in cellular markers of immune activation (IA) is defined as changes in the percentage of cluster of differentiation 4 (CD4) + or cluster of differentiation 8 (CD8)+ T cells that express human leukocyte antigen - antigen D Related (HLA-DR) and cluster of differentiation 38 (CD38). Differences will be tested by using both the Wilcoxon and the t-test.
Time Frame: Between Day 28 of Treatment Phase 1 and Day 28 of Treatment Phase 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 37 | 37
percentage of lymphocytes | 10.00 (5.34) | 9.92 (4.97)
Statistical Analysis 1: Comparison: Rifaximin vs Placebo; We calculated the percentage of total lymphocytes that were expressing activation markers at each time point, and compared the differences in the percentages in the Rifaximin and control groups. We used the Wilcoxon test to detect differences between the differences in percentages in the control and Rifaximin groups; Test type: Superiority; Mean Difference (Net) = 0.7872
Statistical Analysis 2: Comparison: Rifaximin vs Placebo; We calculated the percentage of total lymphocytes that were expressing the activation markers at each time point, and compared the differences in the percentages in the Rifaximin and control groups. We used the T-test to detect differences between the differences in percentages in the control group and Rifaximin groups; Test type: Superiority; p = 0.54, Wilcoxon

5. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: The number of participants with serious and non-serious adverse events that were possibly related to Rifaximin or Placebo as assessed by the Division of Acquired Immune Deficiency Syndrome (AIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0 A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: From baseline until up to approximately 14 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 43 | 45
Participants | 12 | 11

ADVERSE EVENTS:
Time Frame: From baseline until up to approximately 14 weeks.
Description: The Division of Acquired Immune Deficiency Syndrome (AIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, 2004, (Clarification August, 2009) was utilized for grading adverse events. Number of participants affected differ from Participant Flow because it represents the cumulative number of participants analyzed per Arm/Group for this outcome measure.
Arm/Group | Rifaximin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/45
Serious Adverse Events (participants affected / at risk) | 2/43 | 0/45
Other Adverse Events (participants affected / at risk) | 10/43 | 11/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rifaximin (N=43) | Placebo (N=45)
Adenocarcinoma gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rifaximin (N=43) | Placebo (N=45)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2)
Amylase increased (Investigations) | 0 (0) | 1 (1)
Anal examination abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (2)
Bacterial vaginosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood bicarbonate abnormal (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (4)
Blood creatinine increased (Investigations) | 2 (2) | 2 (3)
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Defecation urgency (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Hordeolum (Eye disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 3 (4)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Influenza like illness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Iron deficiency anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lethargy (General disorders) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 1 (2)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Testicular disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2015-07-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT01866826/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2015-07-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT01866826/Prot_SAP_001.pdf